CLINICAL TRIAL: NCT03002207
Title: A Prospective, Comparative Study to Evaluate Effectiveness of Repairing the Defect of Intervertebral Disc With Autologous BMSC and Gelatin Sponge After Microendoscopic Discectomy for Lumbar Disc Herniation
Brief Title: Repairing the Defect of Intervertebral Disc With Autologous BMSC and Gelatin Sponge After Microendoscopic Discectomy for Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhanghao (Other)
Responsible Party: Sponsor-Investigator, Zhanghao, Tianjin Hospital, Tianjin Hospital
Organization: Tianjin Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016(001)
Record Dates: First submitted 2016-12-10; First posted 2016-12-23 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2021-10

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The defect is repaired and sutured (Experimental): Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and they are divided into four groups depend on whether the defect is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge or not and whether the defect is sutured or not. In the first group,the defect of intervertebral disc is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge and sutured.
  Interventions: Device: Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge; Procedure: The defect is sutured
- The defect is repaired but not sutured (Experimental): Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and they are divided into four groups depend on whether the defect is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge or not and whether the defect is sutured or not. In the second group, the defect of intervertebral disc is repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge but not sutured after discectomy.
  Interventions: Device: Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge
- The defect is sutured but not repaired (Experimental): Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and they are divided into four groups depend on whether the defect is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge or not and whether the defect is sutured or not. In the third group, the defect of intervertebral disc is sutured but not repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge after discectomy.
  Interventions: Procedure: The defect is sutured
- The defect is neither sutured nor repaired (No Intervention): Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and they are divided into four groups depend on whether the defect is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge or not and whether the defect is sutured or not. In the four group, the defect of intervertebral disc is neither sutured nor repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge after discectomy.

INTERVENTIONS:
Device: Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge — Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and the defect of intervertebral disc is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge after discectomy.
  Arms: The defect is repaired and sutured; The defect is repaired but not sutured
Procedure: The defect is sutured — Participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and the defect is sutured after discectomy.
  Arms: The defect is repaired and sutured; The defect is sutured but not repaired

SUMMARY:
In this prospective study the investigators seek to evaluate clinical outcomes after repairing the defect of intervertebral disc with autologous BMSC/gelatin sponge during microendoscopic discectomy for participants of lumbar disc herniation.

DETAILED DESCRIPTION:
The participants with lumbar disc herniation diseases are treated by Microendoscopic discectomy, and they are divided into four groups depend on whether the defect is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge or not and whether the defect is sutured or not. In the first group,the defect of intervertebral disc is repaired with Autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge and sutured. In the second group, the defect of intervertebral disc is repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge but not sutured after discectomy. In the third group, the defect of intervertebral disc is sutured but not repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge after discectomy. In the four group, the defect of intervertebral disc is neither sutured nor repaired with autologous Bone Marrow Stem Cell (BMSC)/gelatin sponge after discectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with signs and symptoms of lumbar disc herniation requiring surgical treatment after conservative management;
2. Radiological data on CT/MRI obtained within a period prior to enrollment;
3. Participants give written informed consent before enrollment.

Exclusion Criteria:

1. If participants had an incomplete medical record;
2. Participants had spine tumor, spine infection, previous underwent lumbar surgery, or revision surgery.
3. Participants are taking uninterruptible anticoagulation therapy.
4. Dementia and/or inability to give informed consent.
5. MRI contraindication (e.g. cerebral aneurysm clips, cochlear implants, pacemaker, implanted biostimulators);
6. Pregnancy;
7. Participation in other clinical trial within the last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Oswestry Disability Index(ODI) | Baseline, post-op 3 months, 6 months,12 months
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Changes from baseline in Visual Analogue Scale(VAS) | Baseline, post-op 3 months, 6 months,12 months
  Self reported pain using a 10-point visual analogue scale (0=no pain;10=pain as bad as can be)
Changes from baseline in The Short Form (36) Health Survey(SF-36) | Baseline, post-op 3 months, 6 months,12 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change from Baseline in Magnetic Resonance Classification of Lumbar Intervertebral Disc Degeneration（Pfirrmann classification） | Baseline, post-op 12 months
  The Pfirrmann grading system assesses degenerated intervertebral discs by MRI for the asymmetry in disc structure, distinction of the nucleus and the annulus, signal intensity of intervertebral discs and height of intervertebral discs and assigns grade I to V for disc degeneration。
Change from Baseline in The Height of Disc on MRI Scans | Baseline, post-op 12 months
  Using imaging software, physicians will measure disc height at the treatment discs on the midline T1 sagittal view
Change from Baseline in The Size of Disc Protrusion | Baseline, post-op 12 months
  We will measure the anteroposterior (AP) size of the disc protrusions that required treatment

OTHER OUTCOMES:
The Medical Records | 1 months after hospital discharge
  The Medical Records including operative time、blood loss and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Xinlong Ma, Study Chair — Tianjin Hospital Of Tianjin
Locations (1):
- Tianjin Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakai D, Andersson GB. Stem cell therapy for intervertebral disc regeneration: obstacles and solutions. Nat Rev Rheumatol. 2015 Apr;11(4):243-56. doi: 10.1038/nrrheum.2015.13. Epub 2015 Feb 24. PMID 25708497
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Hernigou P, Poignard A, Beaujean F, Rouard H. Percutaneous autologous bone-marrow grafting for nonunions. Influence of the number and concentration of progenitor cells. J Bone Joint Surg Am. 2005 Jul;87(7):1430-7. doi: 10.2106/JBJS.D.02215. PMID 15995108
- [Derived] Yuan Q, Du L, Xu H, Zhang K, Li Q, Zhang H, Liu Y, Ma X, Xu B. Autologous Mesenchymal Stromal Cells Combined with Gelatin Sponge for Repair Intervertebral Disc Defect after Discectomy: A Preclinical Study in a Goat Model. Front Biosci (Landmark Ed). 2022 Apr 19;27(4):131. doi: 10.31083/j.fbl2704131. PMID 35468690